CLINICAL TRIAL: NCT00527592
Title: A Single Dose Comfort Comparison of Travatan Z in One Eye Versus Xalatan in the Opposite Eye in Patients With Primary Open-Angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: SMA-07-01
Record Dates: First submitted 2007-09-10; First posted 2007-09-11 (Estimated); Results first posted 2010-02-10 (Estimated); Last update posted 2012-05-18 (Estimated); Status verified 2012-05

CONDITIONS: Open-Angle Glaucoma; Ocular Hypertension
Keywords: Comfort
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Travoprost; Latanoprost

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Travoprost (Experimental): Travoprost assigned to one eye, with latanoprost assigned to the fellow eye for intra-individual control. One drop, single dose. The eye, and the order in which the first test medicine was instilled (either travoprost or latanoprost), was randomly assigned.
  Interventions: Drug: Travoprost ophthalmic solution 0.004% with SofZia® preservative system (TRAVATAN Z®)
- Latanoprost (Active Comparator): Latanoprost assigned to one eye, with travoprost assigned to the fellow eye for intra-individual control. One drop, single dose. The eye, and the order in which the first test medicine was instilled (either travoprost or latanoprost), was randomly assigned.
  Interventions: Drug: Latanoprost ophthalmic solution 0.005% (XALATAN®)

INTERVENTIONS:
Drug: Travoprost ophthalmic solution 0.004% with SofZia® preservative system (TRAVATAN Z®) — Ophthalmic solution for the treatment of open-angle glaucoma or ocular hypertension, one drop, single dose. Referred to as travoprost.
  Other Names: TRAVATAN Z®
  Arms: Travoprost
Drug: Latanoprost ophthalmic solution 0.005% (XALATAN®) — Ophthalmic solution for the treatment of open-angle glaucoma or ocular hypertension, one drop, single dose. Referred to as latanoprost.
  Other Names: XALATAN®
  Arms: Latanoprost

SUMMARY:
The purpose of this study is to compare the comfort of Travatan Z in one eye and Xalatan in the opposite eye in patients with primary open-angle glaucoma or ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* Clinical diagnosis of ocular hypertension, primary open-angle, pigment dispersion, or exfoliation glaucoma in both eyes.
* Best corrected visual acuity of 20/200 Snellen or better in each eye.
* Intraocular pressure within protocol-specified range.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Any abnormality preventing reliable applanation tonometry in the study eye(s).
* Any eye conditions or procedures as specified in protocol.
* Progressive retinal or optic nerve disease from any cause.
* Use of contact lenses in the study eye(s).
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2007-05; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from two US glaucoma specialty clinics from 6/8/2007 to 8/13/2008. Eligible patients having a diagnosis of open-angle glaucoma or ocular hypertension in both eyes were enrolled.
Pre-assignment Details: 54 patients were enrolled in the study. Qualified patients ceased prostaglandin use for 3-5 days (wash-out) prior to Visit 2 (randomization).
Groups:
- Travoprost/Latanoprost: Travoprost assigned to one eye, with latanoprost assigned to the fellow eye for intra-individual control.
Period: Overall Study
Arm/Group | Travoprost/Latanoprost
Started | 54
Completed | 54
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Travoprost/Latanoprost
Number analyzed (Participants) | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 17

OUTCOME MEASURES:

1. Primary Outcome: Comfort Immediately After Dosing
Description: Comfort was assessed by the patient and recorded on a scale of 0 to 100, with 0 = perfect comfort and 100 = worse discomfort imaginable.
Time Frame: 5 seconds
Population: Intent to treat: All patients who received test article and completed the trial.
Measure: Mean (Standard Deviation); unit: Units on a scale
Units Other Than Participants: Eyes
Groups:
- Travoprost; Latanoprost: One drop in the study eye, single dose
Arm/Group | Travoprost | Latanoprost
Number analyzed (Participants) | 54 | 54
Number analyzed (Eyes) | 54 | 54
Units on a scale | 7.8 (16.1) | 7.1 (16.2)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study and 14 days post study exit.
Description: This reporting group includes all patients who received test article.
Arm/Group | Travoprost | Latanoprost
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/54
Other Adverse Events (participants affected / at risk) | 0/54 | 0/54

LIMITATIONS AND CAVEATS:
None specified.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor does not guarantee the Investigator's right to publish study results since this is a pilot trial with results intended primarily for internal use. Alcon reserves the right of prior review of any publication or presentation of information related to the study.